CLINICAL TRIAL: NCT04236414
Title: A Phase I, Open-label, Parallel Group Study to Investigate Olaparib Safety and Tolerability, Efficacy and Pharmacokinetics in Paediatric Patients With Solid Tumours
Brief Title: Investigating Safety, Tolerability, Efficacy and PK of Olaparib in Paediatric Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0816C00025; 2023-507904-30-00 (Registry Identifier: CTIS (EU)); 2018-003355-38 (EudraCT Number)
Record Dates: First submitted 2019-11-13; First posted 2020-01-22 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumours
Keywords: Cancer; Malignant cancer; Paediatric population; Olaparib
MeSH Terms: conditions — Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: ≥12 to <18 years (Experimental): Patients will receive a single dose of olaparib on Day 1, followed by initiation of bd continuous dosing from Day 2 onwards. Olaparib tablets should be taken at the same time each day (morning and evening), approximately 12 hours apart with one glass of water. The tablets should be swallowed whole and not chewed, crushed, dissolved or divided. Olaparib tablets can be taken with or without food, with the exception of Day 8 (a PK sampling day) when patients aged ≥3 years old receiving tablets should take olaparib at least 1 hour after food and should refrain from eating for up to 2 hours afterwards.
  Interventions: Drug: Olaparib
- Cohort B: ≥3 to <12 years (Experimental): Patients will receive a single dose of olaparib on Day 1, followed by initiation of bd continuous dosing from Day 2 onwards. Olaparib tablets should be taken at the same time each day (morning and evening), approximately 12 hours apart with one glass of water. The tablets should be swallowed whole and not chewed, crushed, dissolved or divided. Olaparib tablets can be taken with or without food, with the exception of Day 8 (a PK sampling day) when patients aged ≥3 years old receiving tablets should take olaparib at least 1 hour after food and should refrain from eating for up to 2 hours afterwards.
  Interventions: Drug: Olaparib
- Cohort C: ≥6 months to <6 years (Experimental): Patients will receive a single dose of olaparib on Day 1, followed by initiation of bd continuous dosing from Day 2 onwards. Olaparib should be taken at the same time each day (morning and evening), approximately 12 hours apart. Patients in Cohort C will receive a predetermined number of each sprinkle capsule strength (15 and 19.5 mg,) to make up the required dose. Olaparib sprinkle capsules will be administered to the child by the parent/caregiver. Patients in Cohort C are not required to fast including PK sampling days. The dispensed granules should be swallowed whole and not chewed, crushed, dissolved or divided, and should be consumed within 30 minutes of preparation.
  Interventions: Drug: Olaparib
- Signal identification (Experimental): A secondary analysis of response in patients recruited into the signal identification phase will be conducted. Patients included in this analysis must have documented evidence of a deleterious or suspected deleterious germline or tumour HRR gene mutation. A minimum of 10 patients across age and dose cohorts with deleterious or suspected deleterious HRR mutations will be enrolled.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Patients will receive a single dose of olaparib on Day 1, followed by initiation of bd continuous dosing from Day 2 onwards. Olaparib should be taken at the same time each day (morning and evening), approximately 12 hours apart with one glass of water. The tablets should be swallowed whole and not chewed, crushed, dissolved or divided. 25 and 100 mg tablet strengths available for ages ≥3 to <18 years. AAF available for ≥0.5 to <6 years; The AAF is a sprinkle capsule formulation, available in dose strengths of 15 mg and 19.5 mg. The sprinkle capsules contain 1.5 mg granules which are to be dispersed onto a food vehicle prior to dosing.

SUMMARY:
A study to find out whether olaparib is safe and well tolerated when administered to children and adolescents with solid tumours.

DETAILED DESCRIPTION:
A Phase I open-label, multicentre study to determine the RP2D of olaparib monotherapy in the paediatric population, and to evaluate the safety, tolerability, PK, PDx and preliminary efficacy of olaparib monotherapy in paediatric patients from ≥6 months to <18 years of age at enrolment, with relapsed or refractory solid or primary CNS tumours (excluding lymphoid malignancies) for whom there are no standard treatment options. It is anticipated that eligible patients fulfilling all of the inclusion criteria and none of the exclusion criteria, will include but will not be limited to those with osteosarcoma, rhabdomyosarcoma, non-rhabdomyosarcoma soft tissue sarcoma, Ewing Sarcoma, neuroblastoma, medulloblastoma and glioma

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of Informed Consent
* Male and female patients who are ≥6 months to <18 years of age at consent
* Pathologically confirmed relapsed or refractory solid or primary CNS tumours (excluding lymphoid malignancies), with a HRR deficiency/gene mutation, and for whom there are no standard treatment options. Eligible patients may include but not be limited to those with osteosarcoma, rhabdomyosarcoma, non rhabdomyosarcoma soft tissue sarcoma, Ewing Sarcoma, neuroblastoma, medulloblastoma and glioma
* For dose finding phase only: recruitment will be open to all patients with HRR deficiency, based on a local test. For the signal identification phase: recruitment will be open only to patients with documented evidence of a deleterious or suspected deleterious germline or tumour HRR gene mutation that meets the AZ HRR rules
* A formalin fixed, paraffin embedded (FFPE) tumour sample from the primary cancer (all patients) suitable for central HRR testing and a blood sample (patients ≥2 years old) for central germline BRCA testing must be provided for each patient
* For all non-neuroblastoma tumours, patients must have at least 1 radiographical assessable lesion (measurable and/or non-measurable). For neuroblastoma tumours, patients must have radiographical assessable disease with at least 1 lesion (measurable and/or non measurable) OR disease evidenced by uptake of meta-iodobenzylguanidine- (MIBG) or fluorodeoxyglucose positron emission tomography (FDG-PET) scans
* Adequate performance status, organ, and marrow function and adequate weight to obtain blood samples for both safety laboratory assessments and PK analysis.
* Ability to swallow tablets

Key Exclusion Criteria:

* Patients with MDS/AML or with features suggestive of MDS/AML
* Patients unable to swallow orally administered medication
* Unresolved toxicity from previous anticancer therapy
* Unstable or untreated CNS disease (i.e., symptomatic uncontrolled brain metastases or untreated spinal cord compression)
* Previous treatment with a PARP inhibitor, including olaparib
* Receipt of any radiotherapy for cancer treatment (except for palliative reasons) within 30 days prior to first dose of study treatment or receipt of last dose of an approved (marketed) anticancer therapy (chemotherapy, targeted therapy, biologic therapy, monoclonal antibodies, etc) within 21 days prior to the first dose of study treatment
* Concomitant use of known strong or moderate CYP3A inhibitors or concomitant use of known strong or moderate CYP3A inducers
* Whole blood transfusions in the last 120 days prior to screening (packed red blood cells and platelet transfusions are acceptable)

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity [DLTs] | 28 days
  DLT - Dose limiting toxicity
Safety profile | Until 30 days after last dose
  Number of patients with adverse events

SECONDARY OUTCOMES:
Apparent total clearance of the drug from plasma at steady state after oral administration [CLss/F] | The pre-dose sample should be collected within 12±0.5 hours of the Day 7 evening dose of olaparib, prior to the Day 8 morning dose and within 12±1 hours of the Day 28 evening olaparib dose, prior to the Day 29 morning dose.
  Olaparib levels in mcg/mL
Maximum plasma concentration at steady state [Css,max] | The pre-dose sample should be collected within 12±0.5 hours of the Day 7 evening dose of olaparib, prior to the Day 8 morning dose and within 12±1 hours of the Day 28 evening olaparib dose, prior to the Day 29 morning dose.
  Olaparib levels in mcg/mL
Minimum plasma concentration at steady state [Css, min] | The pre-dose sample should be collected within 12±0.5 hours of the Day 7 evening dose of olaparib, prior to the Day 8 morning dose and within 12±1 hours of the Day 28 evening olaparib dose, prior to the Day 29 morning dose.
  Olaparib levels in mcg/mL
Time to maximum plasma concentration at steady state [tss,max] | The pre-dose sample should be collected within 12±0.5 hours of the Day 7 evening dose of olaparib, prior to the Day 8 morning dose and within 12±1 hours of the Day 28 evening olaparib dose, prior to the Day 29 morning dose.
  Olaparib levels in mcg/mL
Area under the curve at steady state [AUCss] | The pre-dose sample should be collected within 12±0.5 hours of the Day 7 evening dose of olaparib, prior to the Day 8 morning dose and within 12±1 hours of the Day 28 evening olaparib dose, prior to the Day 29 morning dose.
  Olaparib levels in mcg/mL
Dose normalised area under the curve at steady state [dose normalised AUCss] | The pre-dose sample should be collected within 12±0.5 hours of the Day 7 evening dose of olaparib, prior to the Day 8 morning dose and within 12±1 hours of the Day 28 evening olaparib dose, prior to the Day 29 morning dose.
  Olaparib levels in mcg/mL
Area under the curve at 0-8 hours [AUC(0-8)] | The pre-dose sample should be collected within 12±0.5 hours of the Day 7 evening dose of olaparib, prior to the Day 8 morning dose and within 12±1 hours of the Day 28 evening olaparib dose, prior to the Day 29 morning dose.
  Olaparib levels in mcg/mL
Area under the curve from zero up to time t [AUC0-t] | The pre-dose sample should be collected within 12±0.5 hours of the Day 7 evening dose of olaparib, prior to the Day 8 morning dose and within 12±1 hours of the Day 28 evening olaparib dose, prior to the Day 29 morning dose.
  Olaparib levels in mcg/mL
Dose normalised maximum plasma concentration at steady state [dose normalised Css,max] | The pre-dose sample should be collected within 12±0.5 hours of the Day 7 evening dose of olaparib, prior to the Day 8 morning dose and within 12±1 hours of the Day 28 evening olaparib dose, prior to the Day 29 morning dose.
  Olaparib levels in mcg/mL
ORR as defined by Investigator-assessed RECIST v1.1, INRC or RANO | Up to 64 months
  ORR - Objective response rate INRC - International Neuroblastoma Response Criteria RECIST - Response Evaluation Criteria in Solid tumours RANO - Response Assessment in Neuro-oncology
DCR as defined by Investigator-assessed RECIST v1.1, INRC or RANO | Up to 64 months
  DCR - Disease control rate INRC - International Neuroblastoma Response Criteria RECIST - Response Evaluation Criteria in Solid tumours RANO - Response Assessment in Neuro-oncology
DoR as defined by Investigator-assessed RECIST v1.1, INRC or RANO | Up to 64 months
  DoR - Duration of response INRC - International Neuroblastoma Response Criteria RECIST - Response Evaluation Criteria in Solid tumours RANO - Response Assessment in Neuro-oncology

CONTACTS AND LOCATIONS:
Overall Officials: Milenkova Tsveta, Study Director — AstraZeneca
Locations (9):
- Research Site, København Ø, Denmark
- France (3):
  - Research Site, Lille
  - Research Site, Toulouse
  - Research Site, Villejuif
- Research Site, Heidelberg, Germany
- Research Site, Seoul, South Korea
- Research Site, Madrid, Spain
- United Kingdom (2):
  - Research Site, Glasgow
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data assessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home